CLINICAL TRIAL: NCT03363607
Title: Comparison Between Digital 3D Printed Transfer Tray Versus Thermoformed Transfer Tray for Indirect Bonding: A Randomized Clinical Trial
Brief Title: Comparison Between Digital 3D Printed Transfer Tray Versus Thermoformed Transfer Tray for Indirect Bonding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Abdelaziz, Resident , MS candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CEBC-CU-2017-11-28
Record Dates: First submitted 2017-11-26; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Orthodontic Indirect Bonding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed transfer tray group (Experimental): Indirect bonding using digital 3D printed transfer tray
  Interventions: Procedure: Digital indirect bonding; Procedure: Intraoral scanning; Procedure: Superimposition and evaluation
- Thermoformed transfer tray group (Active Comparator): Indirect bonding using Thermoformed transfer tray
  Interventions: Procedure: Conventional indirect bonding; Procedure: Intraoral scanning; Procedure: Superimposition and evaluation

INTERVENTIONS:
Procedure: Digital indirect bonding — Indirect bonding of orthodontic attachments using digital 3D printed transfer tray
  Arms: 3D printed transfer tray group
Procedure: Conventional indirect bonding — Indirect bonding of orthodontic attachments using thermoformed transfer tray
  Arms: Thermoformed transfer tray group
Procedure: Intraoral scanning — Intraoral Scanning of the bonded brackets
Procedure: Superimposition and evaluation — superimposition of the brackets' positions before and after bonding and evaluation of the transfer accuracy

SUMMARY:
The study evaluates the accuracy of indirect bonding using 3D printed transfer tray versus thermoformed transfer tray. Half of the brackets will be bonded indirectly using the 3D printed transfer tray and the other half will be bonded indirectly using the thermoformed transfer tray.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking orthodontic treatment with fixed orthodontic appliance.
* Patients with full set of permanent teeth
* Good oral hygiene and periodontal condition.

Exclusion Criteria:

* Patients suffering from any periodontal disease.
* Patients with poor oral hygiene
* Enamel hypoplasia and hypocalcification
* Deep carious lesions / large restorations

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Linear and angular Positioning of the brackets | Immediately after bonding
  To evaluate the transfer accuracy of the brackets by the two transfer trays by measuring the linear and angular differences in the brackets' positions before and after bonding.

SECONDARY OUTCOMES:
Bonding failure of the brackets. | three months
  Evaluation of the bond failure by counting the number of detached brackets immediately and over a three months follow up period.
Chair side time | during the bonding procedure
  To evaluate the chair side time of indirect bonding in each technique